CLINICAL TRIAL: NCT06754735
Title: A Multi-national, Prospective, Randomized, Double Blinded, Placebo-controlled Trial to Evaluate Cyclical Topical Wound Oxygen Therapy (TWO2) in the Treatment of Chronic Venous Leg Ulcers
Brief Title: Trial to Evaluate Cyclical Topical Wound Oxygen Therapy in the Treatment of Chronic Venous Leg Ulcers
Acronym: VaLUe I
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: AOTI Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AOTI
Record Dates: First submitted 2024-12-16; First posted 2025-01-01 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-11

CONDITIONS: Venous Leg Ulcer (VLU)
Keywords: Ulcer, Wound, Randomized, Oxygen, Placebo, Sham, Venous, Compression; Varicose Veins, Venous stasis ulcer; Topical Oxygen
MeSH Terms: conditions — Varicose Ulcer; Ulcer; Wounds and Injuries; Varicose Veins

STUDY DESIGN:
Intervention Model Description: Randomized, Double Blinded, Placebo-controlled Trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The Trial Monitor will be blinded to the participant's allocated intervention.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Topical Wound Oxygen Therapy Device (Active Comparator): Topical Wound Oxygen (TWO2) device in combination with the extremity chamber delivers oxygen and cyclical compression to the wound site. The sealed environment created by the extremity chamber is filled with oxygen for a minimum of 120 minutes, 5 times a week over multilayered compression dressings and a wound contact layer.
  Interventions: Device: Topical Wound Oxygen Therapy
- Sham Control Topical Wound Oxygen (TWO2) device (Sham Comparator): A Sham Control Topical Wound Oxygen (TWO2) device in combination with the extremity chamber that does not deliver oxygen and cyclical compression to the wound site. The sealed environment created by the extremity chamber is filled with room air for a minimum of 120 minutes, 5 times a week over multilayered compression dressings and a wound contact layer.
  Interventions: Device: Sham Control Topical Wound Oxygen

INTERVENTIONS:
Device: Topical Wound Oxygen Therapy — The active intervention is the application of the Topical Wound Oxygen device that supplies cyclical oxygen pressure directly to the wound site within a sealed environment.
  Arms: Topical Wound Oxygen Therapy Device
Device: Sham Control Topical Wound Oxygen — The sham control intervention is the application of Topical Wound Oxygen device that supplies topical room air to the wound site within a sealed environment.
  Arms: Sham Control Topical Wound Oxygen (TWO2) device

SUMMARY:
The purpose of this study is to evaluate the efficacy, safety and economic benefits of Cyclical Pressure Topical Wound Oxygen (TWO2) Therapy in the treatment of venous leg ulcers. Participants will utilize standard of care (SOC) multilayer compression dressings with an inactive wound contact layer. Following a 2-week run-in period with SOC and after meeting all eligibility criteria, subjects will be randomized in a 1:1 ratio with TWO2 therapy or sham control therapy plus SOC. Participants will enter the intervention period of up to 16-weeks, followed by a long-term follow-up period of 52 weeks post randomization.

DETAILED DESCRIPTION:
The full effect of Venous leg ulcers (VLU) on society is poorly understood. While chronic VLU are not considered to have a significant impact on mortality, the burden on patients, caregivers, healthcare systems and related economies cannot be underestimated. VLU affects 2% of the world's population, with 60% progressing to chronic wounds. (1) The reported range of VLU incidence is 0.12 - 1.69% and with a prevalence 0.3 - 1.33%. (2; 3) VLUs are a result of chronic venous insufficiency (CVI) and found to be more prevalent in females than males, with both primary (genetic) and secondary causes that result in valvular incompetence that is further exacerbated by obesity and immobility. (4) With the projected growth of aging and increasingly obese and unhealthy societies, both in the developed and developing world, the anticipated incidence of VLU is expected to rise significantly. (1; 5; 6) It has been well established that the standard of care (SOC) for VLU is the application of conventional compression dressing (CCD), as the successful management of venous hypertension is key to healing VLU. Maintaining a mobile blood flow and delivering oxygen and nutrients to tissues is essential to healing as well as preserving the integrity of skin reducing threat of developing a recurrent VLU.

The role of oxygen in wound healing has been extensively studied. An animal study by Fries et al in 2005 demonstrated that the application of oxygen in partial pressures above those delivered by a well-functioning arterial system, to wounded tissue, resulted in faster healing and more durable tissue. (19) Oxygen is also essential in fighting infection, potentiating the use of antibiotics and upregulating growth factors. (20; 21) A study by Tawfick and Sultan in 2012 demonstrated a significant benefit in healing VLU when both oxygen and cycling compression were employed simultaneously. Utilizing Topical Wound Oxygen (TWO2) therapy™, TWO2 was demonstrated to be superior to SOC, 76% vs 46% healing at 12 weeks (n = 30/65; P < .0001), with low recurrence rates for patients followed up to three years, 6% vs 47%. Further noteworthy results from this study were the reduction of pain, 8 to 3 in 13 days (on a numerical rating scale) and subjects whose wounds were infected with MRSA demonstrated elimination 46% vs 0% at week 5 (P <.001). (22)

All subjects will use the TWO2/Sham device for a minimum of 120 minutes a day in their home (where the infrastructure supports remote therapy), 5 times a week for the treatment phase of up to 16 weeks. Monitoring of the wound will take place with bi-weekly clinic visits to assess safety, compliance, wound progression/deterioration, wound photographs and measurements.

The maximum duration for participation in the trial is 52 weeks (+/- 2 weeks). During the follow-up phase, subjects will receive standard care according to the clinician's recommendation and will be asked not to participate in another wound care trial during this period.

ELIGIBILITY:
Inclusion Criteria:

* Adults ≥ 18 years and able to provide written informed consent
* Patients who have a chronic venous leg ulcer (VLU) below the knee at or above the malleolus determined to be due to underlying venous disease
* Venous reflux ≥ 500 mil sec/superficial or 1 sec/deep or venous mapping after interventions following a vascular procedure
* VLU of ≥ 1.5cm2 and ≤ 50cm2 after debridement at study enrolment i.e. Screening visit
* *Cluster wounds where the sum of the full thickness ulcer area must be ≤ 50cm2
* Study ulcer (current episode of ulceration in case of ulcer recurrence) has been present for at least 6 weeks but no more than 5 years prior to study entry
* The index ulcer has been treated with CCD of at least 30mmHg for ≥ 6 weeks prior to screening.
* Adequate perfusion with Ankle-Brachial Pressure Index (ABPI) of 0.75-1.24 inclusive measured at study entry or within 8 weeks prior to study entry AND TcpO2 > 30mmHg OR Biphasic arterial duplex below the knee OR Toe pressure > 30mmHg OR TBI .6
* Wound size reduction in a 2-week run-in period of ≤ 30%
* Subject understands and is willing to participate in the clinical study and comply with weekly visits and follow up regime
* Subject has read and signed IRB/EC approved ICF before screening procedures commence

Exclusion Criteria:

* • Known allergy to any of the protocol-stipulated treatments, or non-tolerance of multilayer, multicomponent compression therapy

  * Acute thrombophlebitis or Deep Vein Thrombosis (DVT) and within three months preceding study entry
  * Subject awaiting venous ablation or is less than 30 days post ablation
  * Surgery during three months prior to study entry (such as abdominal, gynecological, hip or knee replacement)
  * Wound etiology of uncertain origin or history or prior diagnosis of Systemic Lupus Erythematosus, Burger's Disease, Pyoderma Gangrenosum or other inflammatory ulceration, vasculitis
  * Documented evidence of osteomyelitis on any part of affected limb
  * Index ulcer has exposed bone, muscle and tendon
  * Index ulcer exhibits signs of unmanaged wound infection or severe clinical infection that requires hospitalization or immediate surgical intervention
  * BMI > 45
  * Uncontrolled diabetes: HbA1c > 12% within 60 days of screening
  * Renal dialysis or of screening EGFR less than 30 mg/dl
  * NYHA Class IV
  * Peripheral arterial reconstruction/revascularization on the affected limb within the last 30 days
  * Any medication deemed by the Investigator to potentially interfere with the study treatment (e.g. systemic steroids > 10mg daily dose, immunosuppressive agents).
  * Active systemic treatment for malignancy
  * History of radiation at the ulcer site
  * Subject has received growth factor therapy (e.g., autologous platelet-rich plasma gel, becaplermin, bilayer cell therapy, dermal substitute, extracellular matrix) within 14 days before screening
  * Subject participated in another investigational device, drug or biological trial within four weeks prior to study entry
  * Subject may not be pregnant or breastfeeding at the time of treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 212 (Estimated)
Dates: Start 2025-01-15 (Actual); Primary Completion 2027-06 (Estimated); Study Completion 2028-06 (Estimated)

PRIMARY OUTCOMES:
Incidence of complete wound closure within 16 weeks with the use of Topical Wound Oxygen Therapy (TWO2) | From Baseline to16 weeks
  Percentage incidence of complete wound closure defined as 100% skin re-epithelialization without the need for wound dressing that is confirmed by 2 consecutive study visits 2 weeks apart.

SECONDARY OUTCOMES:
Percentage Area Reduction (PAR) | Baseline, Week 2, 4, 6, 8, 10, 12, 14 up to 16 weeks (± 2 days)
  Change in wound area will be documented bi-weekly by the use of digital photography and wound mapping
Incidence of complete wound closure at 12 weeks | From Baseline to12 weeks
  Incidence of complete wound closure defined as 100% skin re-epithelialization without the need for wound dressing that is confirmed by 2 consecutive study visits 2 weeks apart.
Incidence of complete wound closure at 52 weeks | From week 16 to 52 weeks
  Incidence of complete wound closure defined as 100% skin re-epithelialization without the need for wound dressing that is confirmed by 2 consecutive study visits 2 weeks apart.
Time to complete wound closure | Baseline, Week 2, 4, 6, 8, 10, 12, 14 up to 16 weeks (± 2 days), 20, 26, 52 weeks (± 2 weeks)
  Healing difference over Time will be assessed over a 16-week period
Pain Visual Analog Scale (VAS) score | Baseline weekly up to 16 weeks (±2 days)
  Pain scores documented on a weekly basis measured using a 0-10 Visual Analog Scale (VAS) score, with zero (0) indicating no pain and 10 indicating the worst possible pain.
Incidence of recurrence | From Baseline up to week 16, week 20, 26 (± 1 week), 52 (± 2 weeks)
  Wounds documented as "healed" will be followed for incidence of recurrence. Count of wound recurrences of healed wounds. For healed wounds, VLU recurrence was collected via phone calls and subjects at follow up timelines.
Incidence of Adverse Events at 16 weeks | From Baseline to16 weeks
  Total number of different types of adverse events in participants who reported with any untoward medical event
Incidence of Serious Adverse Events at 16 weeks | From Baseline to16 weeks
  Total number of different types of serious adverse events in participants who reported that:
  * results in death
  * is life-threatening (places the subject at immediate risk of death from the experience as it occurred)
  * results in a persistent or significant disability/incapacity (substantial disruption of one's ability to carry out normal life functions)
  * results in medical or surgical intervention
  * results in or prolongs an existing hospitalization (even if the hospitalization is a precautionary measure for observation)
Incidence of Serious Adverse Events at 52 weeks | From 16 to 52 weeks
  Total number of different types of serious adverse events in participants who reported that:
  * results in death
  * is life-threatening (places the subject at immediate risk of death from the experience as it occurred)
  * results in a persistent or significant disability/incapacity (substantial disruption of one's ability to carry out normal life functions)
  * results in medical or surgical intervention
  * results in or prolongs an existing hospitalization (even if the hospitalization is a precautionary measure for observation)
Change in Venous Clinical Severity Score (VCSS) | From Baseline to 16 weeks
  Mean change in Venous Clinical Severity Score (VCSS) from baseline to week 16. VCSS assesses nine common signs/symptoms of venous disease and each item is scored individually with a minimum score of "0" and maximum score of "3". The individual items are added together to assess change from baseline. Higher scores mean worst outcome.
Elimination of Infection | From Baseline to week 6
  Wound cultures will be taken at the Baseline visit then again at week 6. Wounds defined as "infected" at the baseline visit and "not infection" at weeks 6, are documented as wound infection elimination.
Change in Health-related Quality of Life (Venous Leg Ulcer Quality of life Questionnaire ~ (VLU-QoL-34)) | From Baseline to week 8, up to week 16 (± 2 days)
  Mean difference in change in Venous Leg Ulcer Quality of life Questionnaire ~ (VLU-QoL-34) from baseline to 16 weeks. Crude subscale scores for each group are not shown (each crude subscale is scored 1 to 5 at baseline and 16 weeks); higher mean differences in change from baseline to 16 weeks within groups indicate greater change on the subscales for that group.
Emotional distress | From Baseline to week 8, up to week 16 (± 2 days)
  The emotional distress will be assessed through the total score of the Hospital Anxiety and Depression Scale, comprising both anxiety and depression scales (HADS; Pais-Ribeiro et al., 2007). Scores range between 0 and 42, with higher results indicating higher levels of distress.
Anxiety symptoms | From Baseline to week 8, up to week 16 (± 2 days)
  The anxious symptomatology will be assessed through the Hospital Anxiety and Depression Scale (HADS; Pais-Ribeiro et al., 2007). Scores range between 0 and 21, with higher results indicating higher levels of anxiety symptoms.
Depression | From Baseline to week 8, up to week 16 (± 2 days)
  The depressive symptomatology will be assessed through the Hospital Anxiety and Depression Scale (HADS; Pais-Ribeiro et al., 2007). Scores range between 0 and 21, with higher results indicating higher levels of depression symptoms.
Change in Health-related Quality of Life (EuroQol-5D 3L) | From Baseline to week 8, up to week 16 (± 2 days)
  Mean difference in change measured by EuroQol 5D (EQ5D 3L) from baseline to 16 weeks. Crude health state scores for each group are not shown (health state is scored 0 to 100 at baseline and 16 weeks); higher mean differences in change from baseline to 16 weeks within groups indicate greater change on health state for that group.

CONTACTS AND LOCATIONS:
Overall Officials: Mike Griffiths, DProf, DMS, CRT, FCMI, Study Chair — AOTI Ltd.; Anil Hingorani, MD, Principal Investigator; Wael Tawfick, MB.BCH, MRCSI., Principal Investigator — University of Galway
Locations (1):
- Vascular Institute of New York, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Frykberg RG, Franks PJ, Edmonds M, Brantley JN, Teot L, Wild T, Garoufalis MG, Lee AM, Thompson JA, Reach G, Dove CR, Lachgar K, Grotemeyer D, Renton SC; TWO2 Study Group. A Multinational, Multicenter, Randomized, Double-Blinded, Placebo-Controlled Trial to Evaluate the Efficacy of Cyclical Topical Wound Oxygen (TWO2) Therapy in the Treatment of Chronic Diabetic Foot Ulcers: The TWO2 Study. Diabetes Care. 2020 Mar;43(3):616-624. doi: 10.2337/dc19-0476. Epub 2019 Oct 16. PMID 31619393
- [Background] Tawfick WA, Sultan S. Technical and clinical outcome of topical wound oxygen in comparison to conventional compression dressings in the management of refractory nonhealing venous ulcers. Vasc Endovascular Surg. 2013 Jan;47(1):30-7. doi: 10.1177/1538574412467684. Epub 2012 Dec 5. PMID 23223182
- [Background] Fowkes FG, Evans CJ, Lee AJ. Prevalence and risk factors of chronic venous insufficiency. Angiology. 2001 Aug;52 Suppl 1:S5-15. doi: 10.1177/0003319701052001S02. PMID 11510598
- See also: Related Info — https://aotinc.net/clinical-evidence/